CLINICAL TRIAL: NCT05246033
Title: ACcomplisH China: A Phase 2, Multicenter, Randomized, Placebo-controlled, Dose Escalation Trial Evaluating Safety, Efficacy, and Pharmacokinetics of Multiple Subcutaneous Doses of TransCon CNP Administered Once Weekly in Children With Achondroplasia
Brief Title: A Dose Escalation Trial Evaluating Safety, Efficacy, and Pharmacokinetics of Multiple Subcutaneous Doses of TransCon CNP Administered Once Weekly in Children With Achondroplasia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCC-204
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Achondroplasia
Keywords: Achondroplasia; Dwarfism
MeSH Terms: conditions — Achondroplasia; Dwarfism

STUDY DESIGN:
Intervention Model Description: There are 2 cohorts enrolling 24 subjects who will be randomized to receive either TransCon CNP or Placebo in a 3:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TransCon CNP 50 mcg (Experimental): TransCon CNP 50 mcg CNP/kg or placebo mimicking TransCon CNP 50 mcg delivered once weekly by subcutaneous injection
  Interventions: Drug: TransCon CNP
- TransCon CNP 100 mcg (Experimental): TransCon CNP 100 mcg CNP/kg or placebo mimicking TransCon CNP 100 mcg delivered once weekly by subcutaneous injection
  Interventions: Drug: TransCon CNP
- Placebo (Placebo Comparator): Placebo delivered once weekly by subcutaneous injection
  Interventions: Drug: Placebo for TransCon CNP

INTERVENTIONS:
Drug: TransCon CNP — TransCon CNP drug product is a lyophilized powder in a single-use vial containing either TransCon CNP 3.9 mg CNP-38/vial or TransCon CNP 0.80 mg CNP-38/vial. Prior to use, the lyophilized powder is reconstituted with sterile water for injection and administered by subcutaneous injection via syringe and needle.
  Arms: TransCon CNP 100 mcg; TransCon CNP 50 mcg
Drug: Placebo for TransCon CNP — Weekly subcutaneously injection of placebo.
  Arms: Placebo

SUMMARY:
Purpose of the study:

The main purpose of this study is to determine the safety and evaluate the effect of a once weekly dose of TransCon CNP in prepubertal children with achondroplasia in China.

Study Treatments:

TransCon CNP is an investigational (new) drug, which means that it is currently being tested, and therefore is considered experimental. TransCon CNP is designed to provide a sustained exposure of active CNP by subcutaneous (under the skin) injection once weekly.

The Randomized Period of this study is a double-blinded and placebo-controlled. "Placebo-controlled" means that some participants will receive injections that don't contain any TransCon CNP (placebo injection - no active ingredient). "Double-blinded" means that neither the participant nor the study doctor will know which treatment the participant will be receiving, except in an emergency.

After completion of the Randomized Period the trial participant may be invited to take part of the Open-Label Period of this study.

"Open-label" means that all participants will receive injections that contain TransCon CNP; regardless of which treatment (TransCon CNP or placebo) was assigned during the 52 weeks (1 year) Randomized Period/blinded treatment period. It also means that both the participant and the study doctor will know which treatment, and which dose the participant receives.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of achondroplasia confirmed by genetic testing
2. Age criteria: between ages 2 to 10 years old (inclusive) at Screening Visit
3. Tanner stage 1 breast development for females or testicular volume < 4ml for males at Screening
4. Able to stand without assistance
5. Parent/ legal guardian willing and able to administer subcutaneous injections of study medication
6. Written, signed informed consent of the parent(s) or legal guardian(s) of the participant and written assent of the participant as required by the institutional review board/human research ethics committee/independent ethics committee (IRB/HREC/IEC)

Exclusion Criteria:

1. Clinically significant findings at Screening that:

   * Are expected to require surgical intervention during participation in the trial or
   * Are musculoskeletal in nature, such as Salter-Harris fractures or severe hip pain or
   * Otherwise are considered by the Investigator or Medical Monitor to make a participant unfit to receive investigational medicinal products or undergo trial related procedures
2. Have received any dose of prescription medications intended to affect stature or body proportionality (including human growth hormone) in the 6 months prior to Screening (excluding nutritional supplements)
3. Have received any investigational medicinal product or device intended to affect stature or body proportionality at any time
4. History or presence of injury or disease of the growth plate(s), other than ACH, that affects growth potential of long bones
5. History of any bone-related surgery that affects growth potential of long bones, such as orthopedic reconstructive surgery, including but not limited to:

   * Foramen magnum decompression and laminectomy with full recovery are allowed with minimum of 6 months of bone healing
   * Osteotomy to correct bowing is allowed with 12 months of bone healing
   * Limb-lengthening with full recovery is allowed with a minimum of 12 months of bone healing
   * History of 8 plate epiphysiodesis is allowed, but the plates must have been removed prior to Screening with minimum of 4 weeks of healing
6. Have a growth disorder other than ACH that results in short stature or abnormal growth such as severe achondroplasia with developmental delay and acanthosis nigricans (SADDAN), hypochondroplasia, growth hormone deficiency, Turner syndrome, or pseudoachondroplasia
7. Have a medical condition that could result in short stature or abnormal growth such as inflammatory bowel disease, celiac disease, vitamin D deficiency, untreated hypothyroidism, or poorly controlled diabetes mellitus (HbA1c ≥8.0%), or other diabetic complications. Please note the following allowances:

   * Vitamin D deficiency or insufficiency treated with supplementation is allowed. Vitamin D deficiency is defined as 25(OH)D level <20ng/mL (<49.9 nmol/L), insufficiency is defined as 25(OH)D level <20-30ng/mL (49.92 - 74.86 nmol/L). Participants with Vitamin D deficiency or insufficiency must be on Vitamin D regimen before enrollment
   * Participants with hypothyroidism must be clinically euthyroid for 3 months prior to enrollment and, in the opinion of the Investigator, have achieved any catch-up growth expected from thyroxine replacement
   * Participants with diabetes mellitus must have been on a stable medication regimen for 3 months prior to enrollment (dose adjustments are allowed but addition or discontinuation of medications in this time period is disallowed). In addition to HbA1c <8.0%, any participant with diabetes must have adequate glycemic control in the opinion of the Investigator and Medical Monitor to be considered a good candidate for the trial
8. History or presence of malignant disease, other than basal cell epithelioma/carcinoma or completely resected squamous skin cancer with no recurrence for 12 months per medical records
9. History or presence of the following:

   * Chronic anemia (iron deficiency anemia that is resolved or adequately treated in the Investigator's opinion is allowed)
   * Significant cardiovascular disease per the judgement of the Investigator, such as congenital heart disease (uncomplicated patent ductus arteriosus and atrial or ventricular septal defect with repair are allowed), aortic insufficiency, clinically significant arrhythmias, congestive heart failure with NYHA class II and above or other conditions that impair regulation of blood pressure or heart rate
   * Condition that impacts hemodynamic stability (such as autonomic dysfunction, orthostatic intolerance)
   * Chronic renal insufficiency
   * Chronic or recurrent illness that can affect hydration or volume status. This may include conditions associated with decreased nutritional intake or increased volume loss
   * Bone fracture within 6 months prior to screening (within 2 months for fracture of digits)
   * Any disease or condition that, in the opinion of the Investigator or Medical Monitor, may make the participant unlikely to fully complete the trial, may confound interpretation of trial results, or may present undue risk from receiving investigational product
10. Significant electrocardiogram abnormalities, including evidence of a previous myocardial infarction, left ventricular hypertrophy, flat T waves (particularly in the inferior leads) or more than minor non-specific ST-T wave changes or:

    * QRS >90 milliseconds (msec)
    * QT interval corrected using Fridericia's formula (QTcF) >440 msec
    * PR interval >170 msec
    * Complete right or left bundle branch block
11. Requires, or anticipated to require, chronic (> 4 weeks) or repeated treatment (more than twice/year) with oral corticosteroids during participation in the trial (low and mid-dose inhaled corticosteroids are allowed with Medical Monitor approval. High-dose inhaled corticosteroids are not allowed)
12. Use of medication known to prolong the QT/QTc interval (https://crediblemeds.org/. Note: Only medications on the Known Risk list are excluded, not those on the Possible or Conditional Risk lists). Prior use of such medications is allowed if participant has sufficient wash-out period (minimum 7 days or 5 half-lives, whichever was longer) and a normal QT/QTc interval on ECG.
13. Ongoing treatment with any medication that affects blood pressure or heart rate
14. Known hypersensitivity to the components of the investigational medicinal product (trehalose, tris(hydroxymethyl)aminomethane, succinate and PEG)
15. Any other reason that in the opinion of the Investigator or Medical Monitor would prevent the child from complying with the trial requirements, prevent successful completion of the trial, or prevent successful interpretation of trial data • This could include family situations, comorbid conditions, or medications that might impact safety or be considered confounding

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 52 weeks
  Safety and tolerability of once weekly TransCon CNP treatment or placebo
Annualized height velocity (centimeters/year) at 52 weeks | 52 weeks
  Annualized height velocity measured in centimeters over 52 weeks for TransCon CNP or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Breinholt, Study Director — Ascendis Pharma
Locations (5):
- China (5):
  - Ascendis Pharma Investigational Site, Beijing
  - Ascendis Pharma Investigational Site, Guangzhou
  - Ascendis Pharma Investigational Site, Hangzhou
  - Ascendis Pharma Investigational Site, Shanghai
  - Ascendis Pharma Investigational Site, Wuhan